CLINICAL TRIAL: NCT07261124
Title: Investigation of the Effect of Health Promotion Model Based Oculomotor Exercise Program on Sleep Quality in Elderly Living in a Nursing Home: A Randomized Controlled Trial
Brief Title: Effect of Health Promotion Model-Based Oculomotor Exercise Program on Sleep Quality in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Hande Sabandüzen, PhD Candidate, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IUC_LEE_HS_1
Record Dates: First submitted 2025-11-23; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Sleep Quality; Older Adults (65 Years and Older)
Keywords: sleep quality; health promotion; Eye Movements; nursing; aged
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the experimental or control group using a parallel design. The experimental group will receive a Health Promotion Model-based oculomotor exercise program while the control group will receive no tervention and continue their usual daily activities. Both groups will be evaluated simultaneously at baseline and after the intervention using standardized scales for sleep quality and behavioral change.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants in this group will receive a structured oculomotor exercise program designed according to the Health Promotion Model. The program includes oculomotor exercises performed three times a week and weekly motivational interviewing sessions to enhance self-efficacy and adherence. Sleep quality and behavioral change outcomes will be assessed at baseline and post-intervention.
  Interventions: Behavioral: Oculomotor Exercise Program
- Control Group (No Intervention): Participants in this group will not receive any intervention. They will continue their usual daily activities and will be evaluated using the same measurement tools and time points as the experimental group.

INTERVENTIONS:
Behavioral: Oculomotor Exercise Program — This intervention is a structured oculomotor exercise program based on the Health Promotion Model, developed to improve sleep quality among older adults living in a nursing home. The program focuses on enhancing visual-motor coordination and relaxation through systematic eye movement exercises.
  Participants in the experimental group perform oculomotor exercises three times per week for four consecutive weeks under researcher supervision. The program includes educational support and brief motivational guidance to encourage adherence and consistency. Follow-up sessions are conducted during the following two months to monitor sleep patterns and maintain behavioral improvement.
  This intervention differs from traditional exercise programs by targeting the oculomotor system and incorporating health promotion principles to support better sleep and overall well-being in older adults.
  Arms: Exercise Group

SUMMARY:
The goal of this clinical trial is to investigate the effect of a Health Promotion Model-based oculomotor exercise program on sleep quality among older adults living in a nursing home.

The main questions it aims to answer are:

Does the Health Promotion Model-based oculomotor exercise program improve sleep quality in older adults living in a nursing home? Does participation in the program enhance self-efficacy and promote better health behaviors related to sleep?

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effect of a Health Promotion Model-based oculomotor exercise program on sleep quality among older adults living in a nursing home. Participants in the experimental group will receive an approximately 3-month structured intervention integrating oculomotor exercises and motivational interviewing techniques, while the control group will receive no intervention and continue with their usual daily routines.

The intervention is designed according to the components of the Health Promotion Model, targeting self-efficacy and behavior change processes. During the first meeting, participants complete baseline assessments, including the Personal Information Form, Sleep Beliefs Scale, Stages of Change Inventory, DSM-5 Sleep Disorder Scale, and Pittsburgh Sleep Quality Index (PSQI). Over four weeks, participants in the experimental group perform oculomotor exercises three times a week (Monday, Wednesday, Friday) and attend weekly motivational interviewing sessions focusing on awareness, perceived benefits, self-efficacy, decision balance, empowerment, and commitment to behavior. Weekly DSM-5 Sleep Disorder assessments are also conducted.

Follow-up sessions continue during the second and third months to support maintenance of behavior change, with monthly evaluations using the PSQI and Stages of Change Inventory. Sleep diaries are used throughout to monitor participants' sleep patterns. The primary outcome is sleep quality, and secondary outcomes include self-efficacy and behavioral stage of change.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Residing in the nursing home for at least 6 months
* Scoring 4 or above on the Mini-Cog test
* Pittsburgh Sleep Quality Index (PSQI) score ≥ 5 (indicating poor sleep quality)
* No diagnosis of psychiatric disorders such as depression, bipolar disorder, or schizophrenia
* No diagnosis of serious sleep disorders such as sleep apnea or narcolepsy
* No medical condition causing frequent nocturnal awakenings, such as nocturia
* Not using antipsychotic or other medications that may affect sleep quality
* Having chronic diseases (e.g., diabetes mellitus, hypertension, coronary artery disease) that are controlled with pharmacological treatment
* No communication problems

Exclusion Criteria:

* Older adults unable to perform self-care independently
* Older adults with dizziness or balance problems
* Participants who are hospitalized for any reason during the follow-up or exercise sessions will be excluded from the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | Baseline, 4 weeks, 2 and 3 months after the intervention
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), which evaluates subjective sleep quality, sleep latency, duration, and disturbances over the previous month. Higher scores indicate poorer sleep quality.

SECONDARY OUTCOMES:
Stage of Behavioral Change | Baseline, 4 weeks, 2 and 3 months after the intervention
  Behavioral change related to sleep habits will be assessed using the Stages of Change Inventory. The scale evaluates participants' progression through different stages of adopting and maintaining healthy sleep behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Hande sabandüzen, PhD Candidate, Principal Investigator — İstanbul University-Cerrahpaşa
Locations (1):
- A Nursing home facility in Istanbul, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to privacy and ethical restrictions

REFERENCES:
- See also: Related Info — https://lisansustuegitim.iuc.edu.tr/tr/_